CLINICAL TRIAL: NCT05819190
Title: Efficacy and Safety of Healsea® Hypertonic Nasal Spray 2.7% in the Treatment of Acute Infectious Rhinitis in Adults
Brief Title: Testing the Efficacy in Adults With Cold of HEalsea Rescue*
Acronym: TEACHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lallemand Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LPH-2201
Record Dates: First submitted 2023-03-09; First posted 2023-04-19 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-01

CONDITIONS: Common Cold
Keywords: Acute infectious rhinitis; Rhinosinusitis; Respiratory tract infection; Nasal irrigation
MeSH Terms: conditions — Common Cold; Rhinosinusitis; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healsea Rescue* group (Experimental): Subjects will receive Healsea Rescue* according to its intended use.
  Interventions: Device: Healsea Rescue*
- Placebo group (Placebo Comparator): Subjects will receive Placebo according to identical posology, instructions for use, contraindication, precaution of use and labelling to those of Healsea Rescue.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Healsea Rescue* — Subjects will be administered with Healsea Rescue* by spraying 2 puffs in each nostril 2 times per day during 7 days.
  Arms: Healsea Rescue* group
Device: Placebo — Subjects will be administered with isotonic saline nasal spray indistinguishable from the Healsea Rescue* by spraying 2 puffs in each nostril 2 times per day during 7 days.
  Arms: Placebo group

SUMMARY:
Healsea® Rescue* is a CE-marked class I medical device. This is a saline-based nasal spray supplemented with a natural Symbiofilm™ extract (0.04%) isolated from the marine bacteria. Healsea® Rescue* is indicated in adults for the treatment of symptoms of acute respiratory tract infections, rhinitis or rhinosinusitis, and for reduction of the swelling of the nasal mucosa.

The goal of this clinical trial is to demonstrate that hypertonic saline solution and Symbiofilm™ act in a synergistic manner to alleviate symptoms of the acute rhinitis phase resulting in better efficacy than isotonic saline solution without Symbiofilm™ used as Placebo in adults with early symptoms of common cold / acute infectious rhinitis.

DETAILED DESCRIPTION:
Upper respiratory tract infections (URTIs) and sino-nasal symptoms are very frequent, especially during the fall and the winter. The common cold is caused by a variety of viruses such as human rhinoviruses and influenza viruses. The incidence of acute rhinitis/rhinosinusitis is very high, estimated to occur from 2 to 5 times per year in the average adult. However, the natural course of acute rhinitis in adults is favorable since 75% of persons have a reduction or resolution of symptoms within 7 days. Only 0.5 to 2.0% of subjects develop secondary bacterial sinusitis requiring antibiotic prescription. Bacterial over infections and progression to a chronic state are favoured by the formation of biofilms, which facilitate bacterial growth and persistence as well as reducing antibiotic efficacy. The socioeconomic impact of acute rhinitis is well established: visits to GP, additional prescriptions and over prescription of antibiotics, workdays lost.

Although clinical evidence from well-designed trials is scarce, European and American guidelines for acute rhinosinusitis recommend daily nasal saline irrigation for reduction of the severity of symptoms and for speeding recovery. The exact mechanisms by which nasal irrigation works are not known. However, most of the experts agree that it is primarily a mechanical intervention leading to direct cleansing of the nasal mucosa. Hypertonic saline solutions are generally considered as more effective than isotonic saline solutions in reducing nasal symptoms in the acute phase. Nevertheless, the efficacy of such solution remains moderate.

Healsea® Rescue* is a CE-marked class I medical device. This is a saline-based nasal spray supplemented with a natural Symbiofilm™ extract (0.04%) isolated from the marine bacteria Bacillus licheniformis T14. The nasal solution is hypertonic (NaCl 2.7%). Symbiofilm™ is an exopolysaccharide with emulsifying properties and in vitro antibiofilm activity and detachment properties against various bacterial pathogens. Symbiofilm™ also protects in vitro human nasal epithelial cells viability after Rhinovirus, Adenovirus, Coronavirus OC43 and Flu infection.

The aim of this study is to demonstrate that hypertonic saline solution and Symbiofilm™ act in a synergistic manner to alleviate symptoms of the acute rhinitis phase resulting in better efficacy than isotonic saline solution without Symbiofilm™ used as Placebo.

The study comprises two parts:

- Part 1 (Day1-Day 8): treatment of the acute phase

• with Healsea® Rescue*, 2 puffs in each nostril 2 times per day during 7 days (14 intakes of the investigational device).

or • with isotonic nasal spray (Placebo), 2 puffs in each nostril 2 times per day during 7 days (14 intakes of the Placebo).

- Part 2 (Day 9-Day 13/15): follow-up phase.

The study comprises two visits and one telephone call:

* Visit 1 (V1) at Day 1
* Telephone call at Day 8
* End of study visit (Visit 2, V2) between Day 13 and Day 15.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female subjects >18 years
2. Acute infectious rhinitis/rhinosinusitis for ≤48h before trial entry
3. Symptoms of headache, muscle ache, chilliness, sore throat, blocked nose, runny nose, cough, sneezing with a score ≤9 (according to a self-rated symptom score; scale: 0 → 3 [0: no symptom to 3: severe intensity])
4. At least one of these symptoms: sore throat, runny nose or blocked nose (i.e., with a score ≥1)
5. Willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the information consent form
6. Patient with a smartphone and an internet connection.

Exclusion Criteria:

1. Known hypersensitivity/allergy to any component of the test device
2. Medical history or any current disease that is considered by the investigator as a reason for non-inclusion
3. Severe nasal septum deviation or other condition that could cause nasal obstruction such as the presence of nasal polyps
4. History of nasal or sinus surgery that in the opinion of the investigator may influence symptom scores
5. Antibiotic intake within 2 weeks before screening
6. Systemic or local corticosteroids (nasal route or inhalation) within 4 weeks before screening
7. Antihistamines intake for allergy when treatment was started from less than 4 weeks
8. Chronic decongestant use
9. Recent (within the previous 2 days) intake of a common cold medicine that in the opinion of the investigator may influence symptom score at screening (NSAID, nasal decongestants, cough medicines)
10. Pregnant/Lactating female or absence of efficient contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emil KOLEV, MD, Principal Investigator — DCC Convex Ltd., Sofia, Bulgaria
Locations (1):
- DCC Convex Ltd., Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heikkinen T, Jarvinen A. The common cold. Lancet. 2003 Jan 4;361(9351):51-9. doi: 10.1016/S0140-6736(03)12162-9. PMID 12517470
- [Background] Rosenfeld RM, Piccirillo JF, Chandrasekhar SS, Brook I, Ashok Kumar K, Kramper M, Orlandi RR, Palmer JN, Patel ZM, Peters A, Walsh SA, Corrigan MD. Clinical practice guideline (update): adult sinusitis. Otolaryngol Head Neck Surg. 2015 Apr;152(2 Suppl):S1-S39. doi: 10.1177/0194599815572097. PMID 25832968
- [Background] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- [Background] Rosenfeld RM. CLINICAL PRACTICE. Acute Sinusitis in Adults. N Engl J Med. 2016 Sep 8;375(10):962-70. doi: 10.1056/NEJMcp1601749. No abstract available. PMID 27602668
- [Background] Rabin N, Zheng Y, Opoku-Temeng C, Du Y, Bonsu E, Sintim HO. Biofilm formation mechanisms and targets for developing antibiofilm agents. Future Med Chem. 2015;7(4):493-512. doi: 10.4155/fmc.15.6. PMID 25875875
- [Background] King D, Mitchell B, Williams CP, Spurling GK. Saline nasal irrigation for acute upper respiratory tract infections. Cochrane Database Syst Rev. 2015 Apr 20;2015(4):CD006821. doi: 10.1002/14651858.CD006821.pub3. PMID 25892369
- [Background] Principi N, Esposito S. Nasal Irrigation: An Imprecisely Defined Medical Procedure. Int J Environ Res Public Health. 2017 May 11;14(5):516. doi: 10.3390/ijerph14050516. PMID 28492494
- [Background] Talbot AR, Herr TM, Parsons DS. Mucociliary clearance and buffered hypertonic saline solution. Laryngoscope. 1997 Apr;107(4):500-3. doi: 10.1097/00005537-199704000-00013. PMID 9111380
- [Background] Brown CL, Graham SM. Nasal irrigations: good or bad? Curr Opin Otolaryngol Head Neck Surg. 2004 Feb;12(1):9-13. doi: 10.1097/00020840-200402000-00004. PMID 14712112
- [Background] Rabago D, Zgierska A, Mundt M, Barrett B, Bobula J, Maberry R. Efficacy of daily hypertonic saline nasal irrigation among patients with sinusitis: a randomized controlled trial. J Fam Pract. 2002 Dec;51(12):1049-55. PMID 12540331
- [Background] van Haselen R, Thinesse-Mallwitz M, Maidannyk V, Buskin SL, Weber S, Keller T, Burkart J, Klement P. The Effectiveness and Safety of a Homeopathic Medicinal Product in Pediatric Upper Respiratory Tract Infections With Fever: A Randomized Controlled Trial. Glob Pediatr Health. 2016 Jul 4;3:2333794X16654851. doi: 10.1177/2333794X16654851. eCollection 2016. PMID 27493984
- [Background] Barrett B, Brown RL, Mundt MP, Thomas GR, Barlow SK, Highstrom AD, Bahrainian M. Validation of a short form Wisconsin Upper Respiratory Symptom Survey (WURSS-21). Health Qual Life Outcomes. 2009 Aug 12;7:76. doi: 10.1186/1477-7525-7-76. PMID 19674476
- [Background] Brown RL, Obasi CN, Barrett B. Rasch Analysis of The WURSS-21 Dimensional Validation and Assessment of Invariance. J Lung Pulm Respir Res. 2016;3(2):00076. doi: 10.15406/jlprr.2015.03.00076. Epub 2016 Apr 11. PMID 27812536
- [Background] JACKSON GG, DOWLING HF, SPIESMAN IG, BOAND AV. Transmission of the common cold to volunteers under controlled conditions. I. The common cold as a clinical entity. AMA Arch Intern Med. 1958 Feb;101(2):267-78. doi: 10.1001/archinte.1958.00260140099015. No abstract available. PMID 13497324

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit: 14th December 2022 Last patient last visit: 31 th January 2023 Location: Bulgaria, 1 site
Period: Overall Study
Arm/Group | Healsea Rescue* Group | Placebo Group
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set similar to Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Healsea Rescue* Group | Placebo Group | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (14.0) | 34.4 (13.4) | 35.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 54 | 111
  Male | 43 | 46 | 89
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Bulgaria | 100 | 100 | 200
Total WURSS-21 score at baseline [Mean (Standard Deviation); unit: units on a scale] — Wisconsin Upper Respiratory Symptoms Survey- 21 completed by each subject at baseline.
  Minimal score 0, maximal score 140 (each item is scored from 0 to 7, no symptom/not sick=0 and severe symptom/severely sick =7)
  units on a scale | 37.7 (20.1) | 37.0 (18.2) | 37.4 (19.1)

OUTCOME MEASURES:

1. Primary Outcome: AUC (Area Under Curve) of Wisconsin Upper Respiratory Symptom Survey (WURSS-21) During First 8 Days of Symptoms as Compared Between Both Groups - Full Analysis Set (FAS)
Description: The WURSS-21 questionnaire scores the severity and functional impact of a cold (items 2 to 11 and 12 to 20 respectively) plus 2 items for global severity and global change (items 1 and 21 respectively). Each item is scored from 0 (not sick / Do not have this symptom / Not at all / Very much better) to 7 (severely, severe, severely, very much worse) for global assessment, symptoms, functional impairment and global change respectively. The question 21 is not included in the calculation of the total score of the WURSS-21. The minimum WURSS-21 score is zero (0) and the maximum WURSS-21 score is one hundred forty (140). The questionnaire was completed in a diary once daily in the evening, taking into account the symptoms from the morning to the evening, during Day 2-Day 8 (day of the end of treatment). At Day 1, the WURSS-21 was completed during the visit. After Day 8, it was assessed once daily until the subject feels not sick for two consecutive days.
Time Frame: Treatment period, from Day 1 to Day 8
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Score on a scale*day
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
Score on a scale*day | 135.60 (89.88) | 177.77 (125.40)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; Comparison of the mean AUC of WURSS-21 scores assessed during the first 8 days of the study between both groups - FAS set; Test type: Superiority; p = 0.0192, Wilcoxon (Mann-Whitney)

2. Primary Outcome: AUC (Area Under Curve) of Wisconsin Upper Respiratory Symptom Survey (WURSS-21) During First 8 Days of Symptoms as Compared Between Both Groups - Per Protocol Set (PP)
Description: The WURSS-21 questionnaire scores the severity and functional impact of a cold (items 2 to 11 and 12 to 20 respectively) plus 2 items for global severity and global change (items 1 and 21 respectively). Each item is scored from 0 (not sick / Do not have this symptom / Not at all / Very much better) to 7 (severely, severe, severely, very much worse) for global assessment, symptoms, functional impairment and global change respectively. The question 21 is not included in the calulation of the total score of the WURSS-21. The minimum WURSS-21 score is zero (0) and the maximum WURSS-21 score is one hundred forty (140). The questionnaire was completed in a diary once daily in the evening, taking into account the symptoms from the morning to the evening, during Day 2-Day 8 (day of the end of treatment). At Day 1, the WURSS-21 was completed during the visit. After Day 8, it was assessed once daily until the subject feels not sick for two consecutive days.
Time Frame: Treatment period, from Day 1 to Day 8
Population: Per Protocol Set (PP)
Measure: Mean (Standard Deviation); unit: score on a scale*day
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 58 | 68
score on a scale*day | 122.50 (83.42) | 163.21 (114.00)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; Comparison of the mean AUC of WURSS-21 scores assessed during the first 8 days of the study between both groups - PP set; Test type: Superiority; p = 0.0296, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: AUC of the Symptoms Sub-score (Items 2-11) of the WURSS-21 During First 8 Days
Description: The Symptoms' WURSS-21 questionnaire scores the severity of the cold (items 2 to 11). Each item is scored from 0 (Do not have this symptom) to 7 (Severe). The minimum Symptoms' WURSS-21 score is zero (0) and the maximum is seventy (70). The questionnaire was completed in a diary once daily in the evening, taking into account the symptoms from the morning to the evening, during Day 2-Day 8 (day of the end of treatment). At Day 1, the Symptoms' WURSS-21 was completed during the visit. After Day 8, it was assessed once daily until the subject feels not sick for two consecutive days.
Time Frame: Treatment period, from Day 1 to Day 8
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: score on a sub-scale*day
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
score on a sub-scale*day | 67.11 (43.09) | 87.57 (53.15)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; Test type: Superiority; p = 0.0085, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: AUC of the Quality of Life Sub-score (Items 12-20) of the WURSS-21 During First 8 Days
Description: The Quality-of-Life' WURSS-21 questionnaire scores the impact of the cold on quality of life (items 12 to 20). Each item is scored from 0 (Not at all) to 7 (Severely). The minimum Quality-of-Life' WURSS-21 score is zero (0) and the maximum is sixty three (63). The questionnaire was completed in a diary once daily in the evening, taking into account the symptoms from the morning to the evening, during Day 2-Day 8 (day of the end of treatment). At Day 1, the Symptoms' WURSS-21 was completed during the visit. After Day 8, it was assessed once daily until the subject feels not sick for two consecutive days
Time Frame: Treatment period, from Day 1 to Day 8
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: score on a sub-scale*day
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
score on a sub-scale*day | 54.36 (59.49) | 74.50 (79.15)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; Test type: Superiority; p = 0.0081, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Duration of Cold Symptoms Assessed by Means of the WURSS-21: Duration of Runny Nose
Description: For each item, the duration is defined as the number of symptomatic days between Visit 1 and the first day the subject reports not to have this symptom for two consecutive days.
Time Frame: Through study completion, up to Day 15
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
days | 6.1 (3.1) | 7.2 (3.1)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; Test type: Superiority; p = 0.0050, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Duration of Cold Symptoms Assessed by Means of the WURSS-21: Duration of Plugged Nose
Description: as for outcome 5
Time Frame: Through study completion, up to Day 15
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
days | 5.9 (3.1) | 6.9 (3.2)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; Test type: Superiority; p = 0.0107, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Duration of Cold Symptoms Assessed by Means of the WURSS-21: Duration of Sneezing
Description: as for outcome 5
Time Frame: Through study completion, up to Day 15
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
days | 3.3 (3.4) | 4.3 (3.6)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; Test type: Superiority; p = 0.0424, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Duration of Cold Symptoms Assessed by Means of the WURSS-21: Duration of Sore Throat
Description: as for outcome 5
Time Frame: Through study completion, up to Day 15
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
days | 3.9 (3.7) | 3.9 (3.7)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; 0.05 global significance level (type I error rate); Test type: Superiority; p = 0.430, Wilcoxon (Mann-Whitney) — one sided test

9. Secondary Outcome: Duration of Cold Symptoms Assessed by Means of the WURSS-21: Duration of Cough
Description: as for outcome 5
Time Frame: Through study completion, up to Day 15
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
days | 4.2 (4.3) | 4.3 (3.9)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; 0.05 global significance level (type I error rate); Test type: Superiority; p = 0.339, Wilcoxon (Mann-Whitney); one sided test

10. Secondary Outcome: Duration of Cold Symptoms Assessed by Means of the WURSS-21: Duration of Scratchy Throat
Description: as for outcome 5
Time Frame: Through study completion, up to Day 15
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
days | 4.5 (3.9) | 4.3 (3.8)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; 0.05 global significance level (type I error rate); Test type: Superiority; p = 0.704, Wilcoxon (Mann-Whitney); one sided test

11. Secondary Outcome: Duration of Cold Symptoms Assessed by Means of the WURSS-21: Duration of Hoarseness
Description: as for outcome 5
Time Frame: Through study completion, up to Day 15
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
days | 3.7 (3.9) | 3.9 (3.9)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; 0.05 global significance level (type I error rate); Test type: Superiority; p = 0.298, Wilcoxon (Mann-Whitney); One sided test

12. Secondary Outcome: Duration of Cold Symptoms Assessed by Means of the WURSS-21: Duration of Head Congestion
Description: as for outcome 5
Time Frame: Through study completion, up to Day 15
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
days | 4.7 (4.2) | 3.9 (3.8)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; 0.05 global significance level (type I error rate); Test type: Superiority; p = 0.906, Wilcoxon (Mann-Whitney); one sided test

13. Secondary Outcome: Duration of Cold Symptoms Assessed by Means of the WURSS-21: Duration of Chest Congestion
Description: as for outcome 5
Time Frame: Through study completion, up to Day 15
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
days | 3.1 (3.8) | 3.2 (4.0)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; 0.05 global significance level (type I error rate); Test type: Superiority; p = 0.582, Wilcoxon (Mann-Whitney); one sided test

14. Secondary Outcome: Duration of Cold Symptoms Assessed by Means of the WURSS-21: Duration of Feeling Tired
Description: as for outcome 5
Time Frame: Through study completion, up to Day 15
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
days | 4.7 (3.9) | 4.4 (3.8)
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; 0.05 global significance level (type I error rate); Test type: Superiority; p = 0.743, Wilcoxon (Mann-Whitney); one sided test

15. Secondary Outcome: Cumulative Number of Days of Usual Medication for Common Cold Use
Description: Concomitant treatments (antipyretics, systemic or local mucolytics, decongestants, antitussives, antibiotics) use will be reported in the e-diary by the patient throughout the study, validated by the investigator at the end of study visit before being reported in the e-CRF.
Time Frame: Through study completion, up to Day 15
Population: Full Analysis set
Measure: Number; unit: days
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
days | 7 | 15
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; 0.05 global significance level (type I error rate); Test type: Superiority; p = 0.605, Fisher Exact; One sided test

16. Secondary Outcome: Subject Satisfaction Regarding Ease of Use of the Nasal Spray
Description: At end of study visit (V2) subject satisfaction regarding ease of use will be recorded using a 4-points categorical scale (How would you characterize the use of Healsea® Rescue* nasal spray? 0: not easy ; 1: pretty easy ; 2: easy ; 3: very easy).
Time Frame: Between Day 13 and Day 15
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
Participants
  use not easy | 0 | 1
  use pretty easy | 4 | 3
  use easy | 8 | 9
  use very easy | 88 | 87
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; 0.05 global significance level (type I error rate); Test type: Superiority; p = 1.000, Fisher Exact; one sided test

17. Secondary Outcome: Characterization of Residual Taste by the Subject
Description: At end of study visit (V2) the residual taste after using the spray will be assessed by the subject using a 4-points categorical scale (How would you characterize the residual taste after spraying Healsea® Rescue*?0: not pleasant ; 1: neutral ; 2: pleasant ; 3: very pleasant).
Time Frame: Between Day 13 and Day 15
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
Participants
  residual taste not pleasant | 4 | 3
  residual taste neutral | 59 | 61
  residual taste pleasant | 21 | 21
  residual taste very pleasant | 16 | 15
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; 0.05 global significance level (type I error rate); Test type: Superiority; p = 0.988, Fisher Exact; One sided test

18. Secondary Outcome: Characterization of Cleansing and Moistening of Nasal Mucosa With the Prescribed Treatment by the Subject
Description: At end of study visit (V2) cleansing and moistening of nasal mucosa will be assessed by the subject using a 4-points categorical scale (How would you characterize the cleansing and moistening of nasal mucosa with Healsea® Rescue*?0: no improvement ; 1: slight improvement ; 2: moderate improvement; 3: very clear improvement).
Time Frame: Between Day 13 and Day 15
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healsea Rescue* Group | Placebo Group
Number analyzed (Participants) | 100 | 100
Participants
  no improvement | 3 | 5
  slight improvement | 11 | 11
  moderate improvement | 47 | 37
  very clear improvement | 39 | 47
Statistical Analysis 1: Comparison: Healsea Rescue* Group vs Placebo Group; 0.05 global significance level (type I error rate); Test type: Superiority; p = 0.483, Fisher Exact; one sided test

ADVERSE EVENTS:
Time Frame: throughout the study, up to day 15
Description: Reporting of Adverse events, incidents ( as per EU regulation 2017/745 requirements) and expected side effects
  Incident:
  Means any malfunction or deterioration in the characteristics or performance of a device made available on the market, including use-error due to ergonomic features, as well as any inadequacy in the information supplied by the manufacturer and any undesirable side-effect.
  Expected side effects:
  identified in the manufacturer's labelling
Arm/Group | Healsea Rescue* Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 10/100 | 9/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healsea Rescue* Group (N=100) | Placebo Group (N=100)
pyrexia (General disorders) | 1 (1) | 6 (6) — adverse event
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Incident as per regulation EU 2017/745
nasal disconfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Expected side effect. Did not lead to study or device discontinuation
Application site disconfort (General disorders) | 1 (1) | 0 (0) — Expected side effect. Did not lead to study or device discontinuation
Application site pain (General disorders) | 1 (1) | 0 (0) — Expected side effect. Did not lead to study or device discontinuation
paraesthesia (Nervous system disorders) | 3 (3) | 1 (1) — Expected side effect. Did not lead to study or device discontinuation
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Incident as per regulation EU 2017/745. Did not lead to study or device discontinuation
unpleasant and bitter feeling (General disorders) | 1 (1) | 0 (0) — Incident as per regulation EU 2017/745. Did not lead to study or device discontinuation
nasal cavity pain (General disorders) | 0 (0) | 1 (1) — Incident as per regulation EU 2017/745. Did not lead to study or device discontinuation

LIMITATIONS AND CAVEATS:
There are two limitations of this investigation.

* The symptoms of common cold are known only by subjects. The WURSS-21, a subjective tool for measuring patient reported outcome, was chosen as the most relevant primary endpoint due to lack of easily measurable objective outcome.
* Most subjects had a mild cold with rapid resolution and no complication; it was virtually impossible to assess the impact of using Healsea Rescue* on the intake of acute infectious rhinitis conventional medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT05819190/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT05819190/SAP_001.pdf